CLINICAL TRIAL: NCT02736773
Title: Ridge Preservation With a Low Resorption Xenograft in Posterior Mandible Postextraction Sockets
Brief Title: Xenograft and Posterior Mandibular Socket Filling
Acronym: Flapless
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 9631
Record Dates: First submitted 2016-02-24; First posted 2016-04-13 (Estimated); Last update posted 2019-08-05 (Actual); Status verified 2019-07

CONDITIONS: Xenograft Model
Keywords: Guided Bone; Pre-implant referred; Regeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- xenograft material to slow resorption (Experimental): xenograft material to slow resorption (Bio-Oss®)
  Interventions: Other: xenograft material to slow resorption

INTERVENTIONS:
Other: xenograft material to slow resorption — xenograft material to slow resorption (Bio-Oss®)

SUMMARY:
The aim of this study is to evaluate the volume of madibular bone after placement of a xenograft in a fresh extraction socket in human. The surgery protocol is flapless, and the teeth are mandibular premolars or molars leaving sockets with 4 walls intact or at least 3 walls intact and the buccal wall at 80% . This study will include 35 patients.

DETAILED DESCRIPTION:
Primary objective :

Estimate the percentage of loss of bone volume and the percentage thickness loss of the buccal and palatal cortical for patients who underwent bone volume preservation technology and conservation of the vestibular cortical by guided bone regeneration using a material slow absorption in the molar areas and premolar.

Secondary objectives:

Compare the percentage of loss of bone volume and the percentage loss of thickness of the buccal and palatal cortical patients who underwent a preservation technique, the upgrading data of mandibular posterior region without fillers described in the literature.

Methods :

After tooth extraction of a premolar or molar in mandibular flapless technique, guided bone regeneration is carried out. The cell is filled by a slow absorption material (Xenograft common use). The regeneration space is maintained by a resorbable membrane. To protect the membrane without tissue motion (technical flapless) placing a three-dimensional collagen matrix graft substitute gingival (Muccograft®) will be used. A CBCT preoperative be performed to verify the integrity of cortical and measure the height and width of the residual cavity. caliper measurements at the foot will also be performed during surgery in order to integrate also the thickness of the bone tables and gingival thickness.

After healing of the graft, the pre-implant scan performed at six months postoperatively will measure the height and width of the grafted cell, to compare measurements and evaluate the dynamics of alveolar resorption

ELIGIBILITY:
Inclusion criteria general

* with a unit or avulsion and ROG including 2 adjacent teeth maximum premolars
* aged 18 to 75
* has given its no objection to participate in research Inclusion criteria patient
* Patients can meet the demands of implant treatment (attendance, hygiene)
* Patients showing no indication against-General to surgery

Exclusion criteria patient

• Patient with against-indication for implant treatment. Whether for medical reasons against showing the pre and implant surgery, or local reasons a total loss of vestibular cortical unstabilized periodontal disease or aesthetic cons-indication.

Exclusion criteria general

* Inability to maintain a good level of oral hygiene and good cooperation.
* Higher tobacco consumption has 10cig / day
* Acute dental infection

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2015-12-01 (Actual); Primary Completion 2018-06-01 (Actual); Study Completion 2018-09-01 (Actual)

PRIMARY OUTCOMES:
Cone beam diagnostic examination | Day diagnostic (Day 0)
  Cone beam diagnostic examination: Millimeter measurements will be taken at Day 0.
  This examination is an X-ray technique that uses a cone-shaped radiation beam. The measurements will be made on radiographic examinations
  Mucous measures
  * Vestibular cortical Distance, lingual cortical measured in the middle of the cell
  * Depth of the slot lingual cortical side
  * Depth of the cell vestibular cortical side
  Bone measures
  * Thickness of the lingual cortical measured caliper 2 millimeters under the rim
  * Vestibular cortical thickness measured with calipers 2 millimeters under the rim
  * Depth of the slot lingual cortical side
  * Depth of the cell vestibular cortical side

SECONDARY OUTCOMES:
Cone beam pre implant examination | 5 or 6 months
  Cone beam pre implant examination : millimeter measurements will be taken at 5 or 6 months.
  This examination is an X-ray technique that uses a cone-shaped radiation beam. The measurements will be made on radiographic examinations
  Mucous measures
  * Vestibular cortical Distance, lingual cortical measured in the middle of the cell
  * Depth of the slot lingual cortical side
  * Depth of the cell vestibular cortical side
  Bone measures
  * Thickness of the lingual cortical measured caliper 2 millimeters under the rim
  * Vestibular cortical thickness measured with calipers 2 millimeters under the rim
  * Depth of the slot lingual cortical side
  * Depth of the cell vestibular cortical side
Clinical measures | Day of surgery
  Clinical measures on the day of surgery
  Bone measures
  * Thickness of the lingual cortical measured caliper 2 millimeters under the rim
  * Vestibular cortical thickness measured with calipers 2 millimeters under the rim
  * Cortical vestibular cortical lingual distance, measured in the middle of the cell
  * Depth of the slot lingual cortical side
  * Depth of the cell vestibular cortical side
  Mucous measure:
  * Gum buccal keratinized
  * Keratinized gingiva lingual
  * Cortical vestibular cortical lingual distance measured in the middle of the cell

CONTACTS AND LOCATIONS:
Overall Officials: Philippe BOUSQUET, MCU PH, Principal Investigator — University Hospital, Montpellier
Locations (1):
- UHMontpellier - AHU CSERD, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC